CLINICAL TRIAL: NCT01747863
Title: Prospective Research in Infants With Mild Encephalopathy: the PRIME Study.
Brief Title: Prospective Research in Infants With Mild Encephalopathy
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Brown University (Other); University of Texas Southwestern Medical Center (Other); Wayne State University (Other); Mahidol University (Other); Ohio State University (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Guilherme Sant'Anna, MD, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: PRIME01; 12-108-PED (Other: MUHC)
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Brain Injury; Neonatal Seizure
Keywords: Hypoxic Ischemic encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild NE: Infants with evidence of a perinatal event and NE who do not qualify for therapeutic hypothermia.
  Interventions: Other: Neurologic examination

INTERVENTIONS:
Other: Neurologic examination — Neurologic examination includes: (1) neurologic examination using modify Sarnat score at </= 6 hrs of age, 24 hrs and at discharge home, (2) aEEG at 6 ± 3 hrs of age, (3) Brain MRI before discharge home to 30 days of age.

SUMMARY:
A multicenter observational pilot study will be conducted to determine the natural history of infants with early diagnosis (≤ 6 hrs of age) of mild neonatal encephalopathy (NE) who are not qualified for therapeutic hypothermia. The intervention includes: neurologic examination by using modified Sarnat score at ≤ 6 hrs of age, 24 hrs and before discharge home, amplitude-integrated electroencephalography (aEEG) at 6 ± 3 hrs of age, brain MRI at before discharge home to 30 days of age and follow-up at 18-22 months of age. Primary outcome is the percentage of mild NE infants with evidence of brain injury defined by the presence of at least 1 abnormality of brain MRI, aEEG or neurologic examination in the neonatal period. Secondary outcome is the percentage of brain MRI, aEEG and neurological exam abnormalities, seizure, length of hospital stay, need of gavage feeds or gastrostomy at discharge home, death and long-term outcome.

DETAILED DESCRIPTION:
Globally, an estimated 1.8 to 7.7 infants per 1000 live term births suffer from perinatal asphyxia, which remains an important cause of neonatal encephalopathy (NE) and neurodevelopmental impairment. Over the last six years, several randomized control trials have demonstrated that prolonged and moderate therapeutic hypothermia (TH) reduces the rate of death or disability at 18 months of age among infants who survived. In these trials, infants were eligible if there was evidence of perinatal hypoxia-ischemia and a moderate or severe degree of encephalopathy on neurological evaluation performed at ≤ 6 hrs of age. However, it has been recognized that the level of NE may change over time. Preliminary and unpublished observations from our group indicated that some infants who were not classified as moderate or severe NE had neurological abnormalities at discharge or evidence of brain injury on MRI performed during the neonatal period. Unfortunately, precise data on the outcomes of this specific population is not clear. Since TH is not offered to this population, the outcomes of infants that do not qualify for TH based on neurological evaluation performed ≤ 6 hrs of life requires a more precise investigation.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weight > or = 1800g and gestational age > or = 36 weeks AND
* Admission to neonatal intensive care unit (NICU) for possible hypothermia at < or = 6hr of life

Exclusion Criteria:

* Infants with normal neurological evaluation
* Major congenital abnormalities
* Refusal of informed consent
* Infants who receive passive or active cooling prior to the NICU admission
* Infants that develop seizures or moderate/severe NE within the first 24 hr of life and are initiated on therapeutic hypothermia after 6 hr of life.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with evidence of a perinatal event and NE who do not qualify for therapeutic hypothermia. NE will be defined as the presence of abnormal neurological findings on the modified Sarnat Score performed at ≤ 6 hrs of life. Evidence of a perinatal event will include criteria described in details in the whole body hypothermia trial (NEJM, 2005). The level of NE will be defined by the neurological exam performed by certified neonatologists working at the 6 centers.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Sant'Anna, MD, Principal Investigator — McGill University; Lina Chalak, MD, Principal Investigator — University of Texas; Abbot Laptook, MD, Principal Investigator — Brown University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Chatchay Prempunpong, MD, Principal Investigator — Mahidol University; Sudhin Thayyil, MD, Principal Investigator — Imperial College London; Pablo Sanchez, MD, Principal Investigator — Ohio State University; Pablo Sanchez, MD, Study Director — The Ohio Stage University; Guilherme Sant'Anna, MD, Study Chair — McGill University
Locations (7):
- United States (4):
  - Wayne State University, Detroit, Michigan
  - The Ohio Stage University - Nationwide Children's Hospital, Columbus, Ohio
  - Brown University, Providence, Rhode Island
  - University of Texas Southwestern, Dallas, Texas
- Montreal Children's Hospital, Montreal, Quebec, Canada
- Mahidol University - Ramathibodi Hospital, Bangkok, Thailand
- Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Chalak LF, Adams-Huet B, Sant'Anna G. A Total Sarnat Score in Mild Hypoxic-ischemic Encephalopathy Can Detect Infants at Higher Risk of Disability. J Pediatr. 2019 Nov;214:217-221.e1. doi: 10.1016/j.jpeds.2019.06.026. Epub 2019 Jul 10. PMID 31301853
- [Derived] Prempunpong C, Chalak LF, Garfinkle J, Shah B, Kalra V, Rollins N, Boyle R, Nguyen KA, Mir I, Pappas A, Montaldo P, Thayyil S, Sanchez PJ, Shankaran S, Laptook AR, Sant'Anna G. Prospective research on infants with mild encephalopathy: the PRIME study. J Perinatol. 2018 Jan;38(1):80-85. doi: 10.1038/jp.2017.164. Epub 2017 Nov 2. PMID 29095433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mild NE
Started | 63
Completed | 54
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Mild NE
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Gestational age(weeks)] | 39.4 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants With Evidence of Neurological Dysfunction, Brain Injury and/or Abnormality.
Description: Evidence of neurological dysfunction/injury/abnormality will be defined by any of these 3 criteria, as follows:
  1. MRI = Brain MRI score of pattern of injury (NICHD-NRN) > 0,
  2. aEEG = abnormal background pattern on aEEG (voltage or background pattern) at 6 ± 3 hrs of age.
  3. Any abnormality on the neurological at discharge exam.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Mild NE
Number analyzed (Participants) | 54
Participants | 28

2. Secondary Outcome: Percentage of Infants With Seizures
Description: Development of clinical or electrographic seizures
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 3 days
Reporting Status: Not Posted

3. Secondary Outcome: Length of Hospital Stay
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 3 days
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Infants Who Need Gavage Feeds or Gastrostomy at Discharge Home
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 3 days
Reporting Status: Not Posted

5. Secondary Outcome: Mortality Rate
Description: Death during the hospitalization
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 3 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Long-term Neurodevelopment
Description: Long-term outcomes (18-22 months of age): Severe disability if there is a Bayley III Cognitive score < 70, severe cerebral palsy (CP), defined by the Gross Motor Function Classification System (GMFCS) grade level 3 to 5, blindness or profound hearing loss. Moderate disability will be defined as the Bayley Cognitive score is 70-84 and either seizures, moderate CP (defined by GMFCS grade level 2) or a hearing deficit requiring amplification to understand commands. Mild disability will be defined by a cognitive score 70-84, or a cognitive score ≥ 85 and either presence of mild or moderate CP (GMFCS grade levels 1 or 2), a seizure disorder or hearing loss with or without amplification. Normal will be defined as Bayley III Cognitive score ≥ 85 without any visual or hearing impairment, or CP.
Time Frame: 18-22 months of age
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Mild NE
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No